CLINICAL TRIAL: NCT05261438
Title: Atezolizumab Plus Bevacizumab and Chemotherapy in First-Line Metastatic Nonsquamous NSCLC
Status: Completed | Type: Observational
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, HunanPTH, Hunan Province Tumor Hospital
Other Study IDs: ATRRACT
Record Dates: First submitted 2022-01-22; First posted 2022-03-02 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2019-09

CONDITIONS: Non-squamous NSCLC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — tissue sample and plasma DNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aimed to explore the efficacy of Atezolizumab Plus Bevacizumab and Chemotherapy in First-Line Metastatic Non-squamous NSCLC.

DETAILED DESCRIPTION:
This study aimed to explore the efficacy of Atezolizumab Plus Bevacizumab and Chemotherapy in First-Line Metastatic Non-squamous NSCLC.

ELIGIBILITY:
Inclusion Criteria:

18，Advanced Metastatic Non-squamous NSCLC Treatment Plan is atezolizumab-bevacizumab-carboplatin-paclitaxel

Exclusion Criteria:

Patients with contraindication of chemotherapy Pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced Metastatic Non-squamous Non-small Cell Lung Cancer
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
OS | September 2019- september 2021
  overall survival
PFS | September 2019- september 2021
  progression-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China